CLINICAL TRIAL: NCT03126812
Title: Feasibility Study of Neo-adjuvant Treatment With Carboplatin, Paclitaxel and Pembrolizumab in Primary Stage IV Serous Ovarian Cancer
Brief Title: Neo-adjuvant Pembrolizumab in Primary Stage IV Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N16OPE
Record Dates: First submitted 2016-12-19; First posted 2017-04-24 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer Stage IV; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Primary stage 4; Neo adjuvant
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Carboplatin; Paclitaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carboplatin, paclitaxel, pembrolizumab (Experimental): Carboplatin AUC= 6 paclitaxel 80 mg/m2 Pembrolizumab 200 mg starting cycle 2
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC=6
Drug: Paclitaxel — paclitaxel 80 mg/m2
Drug: Pembrolizumab — 200 mg flat dose, starting cycle 2

SUMMARY:
This is a single arm feasibility study in patients with primary FIGO stage IV serous ovarian, peritoneal, or fallopian tube cancer to evaluate neo-adjuvant + adjuvant pembrolizumab for its capacity to induce and broaden T cell responses against tumor neo-antigens.

DETAILED DESCRIPTION:
Long-term survival in stage IV serous ovarian, peritoneal, and fallopian tube cancer is poor and has not significantly improved over the last decades. Standard treatment consists of debulking surgery and six courses of carboplatin and paclitaxel. Nevertheless, the disease recurs in >90% of women, usually within two years.

Since early observations that the presence of infiltrating T cells is associated with improved outcome, ovarian cancer is linked to a potential benefit of immunotherapy.10 More recently, T cell checkpoint blockade with anti-PD1 and anti-PDL1 have shown promising activity in platinum resistant ovarian cancer with objective and durable responses in 10-20% of patients. This finding raises the question whether anti-PD1 could also play a role in first line treatment of ovarian cancer.

To fully use the power of T cell checkpoint inhibition, sufficient TCR stimulation is required. Importantly, the amount of antigen that can provide this signal will correlate with tumor load, and because of this adjuvant immunotherapy may work most efficiently, when initiated prior to surgery. In addition, we postulate that antigen retrieval will increase after induction treatment with cytotoxic therapy.

To address these questions, we propose a feasibility study in patients with FIGO stage IV serous ovarian, peritoneal, or fallopian tube cancer in which we evaluate pembrolizumab added to standard treatment for its capacity to induce and broaden T cell responses against neo-antigens.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for the trial.
* Diagnosis of primary stage IV high-grade serous ovarian, peritoneal, or fallopian tube cancer.
* Age >= 18 years on day of signing informed consent.
* Willing and able to provide three tumor biopsies (1 FFPE, 2 fresh frozen) prior to start of treatment
* Performance status of 0 or 1 on the ECOG Performance Scale.
* Adequate organ function as defined in Table 1 of the protocol
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Exclusion Criteria:

* Previously received treatment for ovarian, peritoneal, or fallopian tube cancer.

  * Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
  * Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Known additional malignancy, unless treated with curative intent without chemotherapy at least five years ago. In situ cancers, basal cell carcinoma of the skin or squamous cell carcinoma of the skin that have undergone potentially curative therapy within the past five years may also be eligible.
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* A diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* A known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Number of T-cells in peripheral blood | up to week 52
  determine the number of T cells in peripheral blood samples and tissue samples

SECONDARY OUTCOMES:
Toxicity; Incidence of toxicity, graded according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4.0 | up to 30 days after end of treatment
  Toxicity will be analyzed in patients who have received at least one administration of pembrolizumab.
Response Rate | at week 12, debulking surgery
  number of patients with no viable invasive tumor left in the resection specimen
Response rate according to RECIST | at week 3 and 6
  Number of patients with partial or complete response according to RECIST

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
to be determinated